CLINICAL TRIAL: NCT06818383
Title: Four-year Follow-up in Rezum Therapy of Small Prostates in Comparison with Large Prostates. a Prospective Trial
Brief Title: Comparative Study Between Rezum Therapy in Small and Large Prostates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: khaled Abdelsattar Gad Ibrahim (Other)
Responsible Party: Sponsor-Investigator, khaled Abdelsattar Gad Ibrahim, consultatnt doctor, Armed Forces College of Medicine, Cairo, Egypt
Organization: Armed Forces College of Medicine, Cairo, Egypt (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rezum therapy in prostate
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Prostate Hyperplasia
Keywords: Rezum; LUTS
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BPH patients have small prostates treated with Rezum (Active Comparator): Patients aged 45-75 years with prostate volumes of 50-80 ml, sexually active, and have severe LUTS treated with Rezum procedure
  Interventions: Device: Rezum therapy
- BPH patients have large prostates treated with Rezum (Active Comparator): Patients aged 45-75 years with prostate volumes of 80-120 ml, sexually active, and have severe LUTS treated with Rezum procedure
  Interventions: Device: Rezum therapy

INTERVENTIONS:
Device: Rezum therapy — minimal invasive technique for treating BPH

SUMMARY:
The investigators aimed to compare the efficacy and safety of Rezūm therapy for the management of benign prostatic hyperplasia (BPH) in small and large prostates.

DETAILED DESCRIPTION:
For decades, Transurethral resection of the prostate (TURP) was the gold standard surgical intervention for small and moderate prostates, however it has high morbidity and prolonged hospital stay Rezūm is a radiofrequency made water vapour thermal treatment. It has recently been added to the international guidelines as a choice for medical treatment resistant lower urinary tract symptoms (LUTS). The AUA and Canadian Urological Association (CUA) guidelines now add water vapour therapy as a treatment option for BPH patients with small prostate size <80 gm and for those wishing to maintain antegrade ejaculation. While investigators still offer no clear recommendation to Rezūm use for those with large prostates.

ELIGIBILITY:
Inclusion Criteria:

1. prostate size 45-75 gm
2. sexually active
3. mod - sever LUTS
4. Q max < 15
5. IPSS > 15
6. failed medical treatment with alpha blockers

Exclusion Criteria:

1. neurogenic bladder
2. urethral stricture
3. UB stones
4. cancer prostate

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — because the prostates in males only
Enrollment: 178 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
The Maximum Urinary flow rate (Qmax) | for each case in both groups the investigator assess Qmax at 3, 12, 24, 36 and 48 months after procedures through study completion, an average of 4 years]
  Measurement of The Maximum Urinary flow rate (Qmax) in both groups After 3, 12, 24, 36 and 48 months of operation, the procedure is performed. Qmax is measured by (ml/sec) Normal values are described as a Qmax above 15 ml/sec and below 10 ml/sec is considered abnormal
The Quality of Life (QoL) | for each case in both groups the investigator assess QoLat 3, 12, 24, 36 and 48 months after procedures through study completion, an average of 4 years]
  Measurement of The Quality of Life (QoL) in both groups After 3, 12, 24, 36 and 48 months of operation, the questioner is performed. Minimum :0 means delighted / Maximum : 5 means unhappy
The Prostatic specific antigen (PSA) | for each case in both groups the investigator measures PSA at 3, 12, and 24, 36 and 48 months after procedures through study completion, an average of 4 years
  Concentration of The Prostatic specific antigen (PSA) in both groups after 3, 12, 24, 36 and 48 months of operation, the procedure is performed. PSA is measured by ng/ml PSA levels of 4.0 ng/ mL and lower were considered
The International Prostate Symptom score (IPSS) | for each case in both groups the investigator assess IPSS at 3, 12, 24, 36 and 48 months after procedures through study completion, an average of 4 years
  Measurement of The International Prostate Symptom score (IPSS) in both groups After 3, 12, 24, 36 and 48 months of operation, the questioner is performed. Minimum :0 / Maximum : 35 Total score: 0-7 Mildly symptomatic; 8-19 moderately symptomatic; 20-35 severely symptomatic
The International Index of Erectile Function (IIEF) | for each case in both groups the investigator assess IIEF at 3, 12, 24, 36 and 48 months after procedures through study completion, an average of 4 years
  Measurement of The International Index of Erectile Function (IIEF) in both groups After 3, 12, 24, 36 and 48 months of operation, the questioner is performed. The IIEF-5 score is the sum of the ordinal responses to the 5 items.
The Prostate size | for each case in both groups the investigator assess prostate size at 12, 24, 36 and 48 months after procedures through study completion, an average of 4 years
  the prostate size was measured by grams by Trans-rectal ultra sound
The operative time | for each case in both groups the investigator assess the time of operation from induction of anaesthesia till the end of the operation through study completion, an average of 4 years
  the operative time was measured by minutes in both groups.
Incidence of The catheter duration post operative | for each case in both groups the investigator assess the catheter duration from the end of the operation till removal through study completion, an average of 4 years
  The catheter duration was measured by days in both groups
Post operative hospital stay time | for each case in both groups the investigator assess the hospital time from the day of admission of the patient in hospital to do intervention till discharge from hospital through study completion, an average of 4 years
  the Post operative hospital stay time was measured by hours in both groups.
Post operative residual urine (PVR) | for each case in both groups the investigator assess prostate size at 3, 12, 24, 36 and 48 months after procedures through study completion, an average of 4 years
  PVR was measured by ml by pelvi abdominal ultra sound in both groups. Normal ranges are below 150 ml of urine.

SECONDARY OUTCOMES:
Incidence of complications | through four years
  For each case in both groups the investigator assess the safety using incidence of complications by The Clavien-Dindo system

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Samir Salem, MD, Study Chair
Locations (1):
- The Armed Forces College of Medicine (AFCM), Cairo, Nozha, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bole R, Gopalakrishna A, Kuang R, Alamiri J, Yang DY, Helo S, Ziegelmann MJ, Kohler TS. Comparative Postoperative Outcomes of Rezum Prostate Ablation in Patients with Large Versus Small Glands. J Endourol. 2020 Jul;34(7):778-781. doi: 10.1089/end.2020.0177. Epub 2020 Jun 12. PMID 32408768
- [Background] McVary KT, Rogers T, Roehrborn CG. Rezum Water Vapor Thermal Therapy for Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia: 4-Year Results From Randomized Controlled Study. Urology. 2019 Apr;126:171-179. doi: 10.1016/j.urology.2018.12.041. Epub 2019 Jan 21. PMID 30677455
- [Background] Dixon CM, Cedano ER, Pacik D, Vit V, Varga G, Wagrell L, Larson TR, Mynderse LA. Two-year results after convective radiofrequency water vapor thermal therapy of symptomatic benign prostatic hyperplasia. Res Rep Urol. 2016 Nov 21;8:207-216. doi: 10.2147/RRU.S119596. eCollection 2016. PMID 27921028
- See also: efficay of Rezum tehrapy in large prostates — https://pmc.ncbi.nlm.nih.gov/articles/PMC7779102/